CLINICAL TRIAL: NCT04874181
Title: A Proof Of Concept Single Arm Study To Use Virtual Reality in Rehabilitation of Stroke Patients in Neuro Intensive Care Unit in Tan Tock Seng Hospital
Brief Title: Use of Virtual Reality Game in Rehabilitation of Stroke Patients in Tan Tock Seng Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020/00143
Record Dates: First submitted 2020-07-05; First posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2020-07

CONDITIONS: Stroke, Acute
Keywords: virtual reality; Silverfit 3D; rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Single Arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Silverfit 3D (Experimental): The subject will use SIlverfit 3D for rehabilitation of his/her shoulder/knee strength post stroke.
  Interventions: Device: Silverfit 3D

INTERVENTIONS:
Device: Silverfit 3D — Virtual reality game used for rehabilitation of stroke patients

SUMMARY:
Use of SIlverfit 3d to aid in rehab of stroke patients focusing on their shoulder and knee strength

DETAILED DESCRIPTION:
Either 1 of 3 physiotherapists will recruit the patient from NICU if the GCS is 14 - 15. Silverfit 3D will then be used for 20 minutes each day to train the knee and arm strength until the patient's discharge from ICU. Baseline muscle strength will be measured and graded by the physiotherapist using Medical Research Council grading then followed up by the same physiotherapist on discharge from ICU and on discharge from hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients 21 - 90 years old
* Diagnosis of stroke of pure motor/sensory type affecting the limbs, all levels of severity and at all stages post stroke, defined by the WHO as "a syndrome of rapidly developing symptoms and signs of focal, and at times global, loss of cerebral function lasting more than 24 hours or leading to death with no apparent cause other than that of vascular origin" (WHO 1989), diagnosed by imaging or neurological examination
* GCS 14 - 15
* RASS -1 to +1
* Blood pressure within 20% of patient's baseline
* Muscle power at least 2 out of 5 on the affected side, as assessed by the physiotherapist or clinician

Exclusion Criteria:

* Age less than 21 or more than 90 years old
* Neurological instability
* Poor prognosis/expected withdrawal of treatment/palliative care patient
* Visual loss/hearing loss
* Active delirium with inability to cooperate as determined by CAM-ICU positivity
* Severe cognitive impairment/dementia
* Haemodynamic instability

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-04-13 (Actual)

PRIMARY OUTCOMES:
To estimate an improvement in muscle strength using the Medical Research Council (MRC) grading following the intervention. | 3 months
  Use of MRC grade to estimate improvement in muscle strength by a group of trained physiotherapists before, during and after the use of virtual reality equipment.
estimate how much a patient can do compared to his/her baseline in terms of ability to stand/ambulation/reaching out for objects based on the physiotherapist who first saw the patient. | 3 months
  Patients will be interviewed on admission by the physiotherapist to find out his/her baseline activities of daily living/strength and limb power. Physiotherapists will assess the patient again on day of discharge to find out how much the patient is able to return to his/her baseline post stroke. This is a descriptive outcome measure as it is only measured by 1 physiotherapist who has seen the patient on admission and then on discharge from hospital.
increase frequency and intensity of rehab activities in stroke patients | 6 months
  To increase frequency of rehab activities in patients in terms of percentage of patients who can do, time of each exercise

SECONDARY OUTCOMES:
reduce length of stay in ICU | 3 months
  Reduce length of stay in ICU

CONTACTS AND LOCATIONS:
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No